CLINICAL TRIAL: NCT03162757
Title: Comparison of Ultrasound-guided Central Venous Catherterization Via the Lower Internal Jugular Vein or the Subclavian Vein
Acronym: JI vs SC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Local/2016/CR-02; 2016-A01400-51 (Other: ANSM)
Record Dates: First submitted 2017-05-12; First posted 2017-05-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2019-01

CONDITIONS: Central Venous Access
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subclavian vein access (Experimental)
  Interventions: Procedure: Central venous catheterization
- Internal jugular vein access (Experimental)
  Interventions: Procedure: Central venous catheterization

INTERVENTIONS:
Procedure: Central venous catheterization — Central venous catheterization via either internal jugular vein or subclavian vein up to a maximum of two attempts.

SUMMARY:
The aim of this pilot study is to establish the success rate of catheterization of the lower jugular vein and the subclavian vein under ultrasound guidance in real time. The purpose is to compare the two techniques and to determine the best design for a full study (superiority, non-inferiority). This is a 2-arm randomized control study. The randomization ensures the comparability of the groups and allows evaluation of the feasibility and potential bias for further comparative studies.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been, or will be, informed as soon as their state of health allows them to be entered into the study of its objectives, constraints and the patient's rights
* The patient have given their free and informed consent and signed the consent form
* The patient must be insured or a beneficiary of a health insurance plan
* The patient is over 18 years old
* The patient needs a venous catheter in the superior vena cava

Exclusion Criteria:

* The patient is already participating in another interventional study that could influence the results of this study
* The patient has participated in another interventional study within the previous 3 months that could influence the results of this study
* The patient is in a period of exclusion determined by a previous study
* The patient is under judicial protection or is an adult under guardianship
* The patient refuses to sign the consent form
* Non-echogenic patient
* Moribund patient
* The patient has a contra-indication to one or other of the approaches: infection of the insertion zone, known thrombosis, severely dyspneic
* Patient has severe coagulation problems: PT<40%, platelets<50 000 and curable anticoagulation with antiXa > 0.5 or INR>3.
* Patient has a congenital or acquired deformation at the entry site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Successful placement catheter from a maximum of two attempts | During procedure
  Binary yes/no

SECONDARY OUTCOMES:
Pneumothorax | 1 day
  binary yes/no
arterial puncture | within 1 hour
  binary yes/no
failure | within 1 hour
  binary yes/no
arrhythmia | within 1 hour
  binary yes/no
abberant placement of catheter | 1 day
  binary yes/no
catheter infection | at removal of catheter; on average 6.5 days
  binary yes/no
catheter colonization | at removal of catheter; on average 6.5 days
  binary yes/no
mediastinal hematoma | 1 day
  binary yes/no
thrombosis | until removal of catheter; on average 6.5 days
  binary yes/no
success at first attempt | within 1 hour
  yes/no
time between puncture until insertion of guide | within 1 hour
  measure in seconds
clinical variables associated with failure of the techniques | within 24 hours
number of dressings | over length of hospitalization; maximum 40 days
  per day
nurse-rated satisfaction at each dressing replacement | over length of hospitalization; maximum 40 days
  score 0-10
haemothorax | 1 day
  binary yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fournil C, Boulet N, Bastide S, Louart B, Ambert A, Boutin C, Lefrant JY, Muller L, Roger C. High success rates of ultrasound-guided distal internal jugular vein and axillary vein approaches for central venous catheterization: A randomized controlled open-label pilot trial. J Clin Ultrasound. 2023 Jan;51(1):158-166. doi: 10.1002/jcu.23383. Epub 2022 Nov 17. PMID 36385459